CLINICAL TRIAL: NCT06678464
Title: An Exploratory, Prospective, Open-label, Randomized, Three-arm, Single-centre, Safety, Efficacy and In-use Tolerability Study of the Three Different Test Products in Healthy Adult Human Subjects With Dry and Sensitive Skin.
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Test Products in Healthy Adult Human Subjects With Dry and Sensitive Skin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Glowderma Lab Private Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NB240044-GL
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dry and Sensitive Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moiz MM (Experimental): 1. Mode of Usage: After cleansing, apply liberally onto the skin and gently massage until fully absorbed.
  Manufactured By: Dermalogics Marketed By: Glowderma Lab Private Limited Frequency: Twice a Day Route of Administration: Topical
  Interventions: Other: Moiz MM
- Moiz XL (Experimental): Mode of Usage: After cleansing, apply liberally onto the skin and gently massage until fully absorbed.
  Manufactured By: Dermalogics Marketed By: Glowderma Lab Private Limited Frequency: Twice a Day Route of Administration: Topical
  Interventions: Other: Moiz XL
- Moiz LMF 48 (Experimental): Mode of Usage: After cleansing, apply liberally onto the skin and gently massage until fully absorbed.
  Manufactured By: Dermalogics Marketed By: Glowderma Lab Private Limited Frequency: Twice a Day or as often as needed Route of Administration: Topical
  Interventions: Other: Moiz LMF 48

INTERVENTIONS:
Other: Moiz MM — Mode of Usage: After cleansing, apply liberally onto the skin and gently massage until fully absorbed.
  Manufactured By: Dermalogics Marketed By: Glowderma Lab Private Limited Frequency: Twice a Day Route of Administration: Topical
  Arms: Moiz MM
Other: Moiz XL — Mode of Usage: After cleansing, apply liberally onto the skin and gently massage until fully absorbed.
  Manufactured By: Dermalogics Marketed By: Glowderma Lab Private Limited Frequency: Twice a Day Route of Administration: Topical
  Arms: Moiz XL
Other: Moiz LMF 48 — Mode of Usage: After cleansing, apply liberally onto the skin and gently massage until fully absorbed.
  Manufactured By: Dermalogics Marketed By: Glowderma Lab Private Limited Frequency: Twice a Day or as often as needed Route of Administration: Topical
  Arms: Moiz LMF 48

SUMMARY:
An exploratory, prospective, open-label, randomized, three-arm, single-centre, safety, efficacy and in-use tolerability study of the three different test products in healthy adult human subjects with dry and sensitive skin.

This exploratory, prospective, open-label, randomized, three-arm, single-centre, safety, efficacy and in-use tolerability study of the three different test products in healthy adult human subjects with dry and sensitive skin.

DETAILED DESCRIPTION:
A total of up to 84 (28 subjects/arm) healthy male and non-pregnant | non-lactating female with equal distribution of dry and sensitive skin (1:1) with an age of 18-55 years will be enrolled to complete the 75 subjects (25 subjects/arm) the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called telephonically by the recruiting department prior to the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day.

Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluation, On Site Product Usage, Post Usage Evaluation

* Visit 02 (Day 08 +2 Days): Evaluations, Product usage period
* Visit 03 (Day 30 +2 Days): Product Usage Period, Evaluations
* Visit 04 (Day 60 +2 Days): Evaluations, End of Study

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18 to 55 years (both inclusive) at the time of consent. 2) Sex: Healthy male and non-pregnant/non-lactating females. 3) Females of childbearing potential must have a self-reported negative pregnancy test.

  4) Subject are generally in good health. 5) Subject with dry and sensitive skin at a time of screening. (Dermatological Assessment) 6) Subjects forearm must be free of cuts, tattoos, scratches, abrasions, scars, uneven skin tone, sunburn, excessive tan, excessive hair or open wounds on or near the test sites.

  7) Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.

  8) If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.

  9) Subjects are willing to give written informed consent and are willing to come for regular follow up.

  10) Subjects who commit not to use medicated skincare products other than the test product for the entire duration of the study.

  11) Subject who have not participated in a similar investigation in the past three months.

  12) Willing to use test product throughout the study period.

Exclusion Criteria:

* 1) History of any dermatological condition of the skin diseases. 2) Subject with present condition of allergic response to any cosmetic product. 3) Subject having allergic response to the ink. 4) any areas of broken/chapped/cut/irritated/scraped skin. 5) Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.

  6) Subject having acne of severe incidence (presence of nodules, cysts or numerous pustules) which requires pharmaceutical or cosmeceuticals, herbal treatment.

  7) Subjects who have applied topical treatment for at least 4 weeks and any systemic treatment for at least 3 months, before they participated in the study.

  8) History of alcohol or drug addiction. 9) Subjects using other marketed products during the study period. 10) Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.

  11) Pregnant or breastfeeding or planning to become pregnant during the study period.

  12) History of chronic illness which may influence the cutaneous state. 13) Subjects participating in other similar cosmetics, devices or therapeutic trials or skincare products within the last four weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of the test products in terms of change in skin hydration | before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Instrumental evaluation by Corneometer CM 825
To assess the effectiveness of the test products in terms of change in DASI score | before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Using DASI Score where 0 is absent 4 is extreme
To assess the effectiveness of the test products in terms of change in overall dry skin score (ODS) | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Using scoring scale where 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in PGA score | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Scoring scale where 0 is none and 8 is extreme
To assess the effectiveness of test products in terms of change in skin barrier function | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Instrumental Evaluation by Tewameter TM Hex
To assess the effectiveness of the test products in terms of change in skin roughness | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Using Scoring Scale 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in skin scaliness | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Using Scoring Scale 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in skin smoothness | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Using Scoring Scale 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in skin wrinkles | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  Using Scoring Scale 0 is absent and 4 is extreme

SECONDARY OUTCOMES:
To assess the effectiveness of the test product in terms of change in desquamation index | before usage of the test products on Day 01 and after usage of the test products at T20 mins on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days)
  using instrumental evaluation of VISIOSCAN VC 20 Plus though Corneofix® F 20

OTHER OUTCOMES:
To assess the effectiveness of the test products in terms of change in visual assessment of skin dryness | before usage of the test products on Day 01, after usage of the test products at T20 min on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days).
  Using a scoring scale where 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in visual assessment of skin smoothness | before usage of the test products on Day 01, after usage of the test products at T20 min on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days).
  Using a scoring scale where 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in visual assessment of skin roughness | before usage of the test products on Day 01, after usage of the test products at T20 min on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days).
  Using a scoring scale where 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in visual assessment of skin redness | before usage of the test products on Day 01, after usage of the test products at T20 min on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days).
  Using a scoring scale where 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in visual assessment of skin itchiness | before usage of the test products on Day 01, after usage of the test products at T20 min on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days).
  Using a scoring scale where 0 is absent and 4 is extreme
To assess the effectiveness of the test products in terms of change in visual assessment of skin scaliness. | before usage of the test products on Day 01, after usage of the test products at T20 min on Day 01, Day 08 (+2 Days), Day 30 (+2 Days) and Day 60 (+2 Days).
  Using a scoring scale where 0 is absent and 4 is extreme

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India